CLINICAL TRIAL: NCT05052645
Title: Auricular Acupuncture in the Treatment of Neuropathic Pain: A Randomized Controlled Trial
Brief Title: Ear Acupuncture for Neuropathic Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigators have limited availability
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tony Y. Chon, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-010454
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (No Intervention): Subjects will receive standard of care neuropathic pain treatment without acupuncture.
- Acupuncture Treatment Group (Experimental): Subjects will receive acupuncture treatment in addition to to the standard of care neuropathic pain treatment.
  Interventions: Procedure: Auricular acupuncture

INTERVENTIONS:
Procedure: Auricular acupuncture — Placement of acupuncture needles in specific points on the ear in two consecutive treatments spaced 7 days apart.
  Arms: Acupuncture Treatment Group

SUMMARY:
The purpose of this study is to gather information on the effectiveness of auricular acupuncture (i.e., the placement of acupuncture needles in specific points on the ear) in reducing pain and improving quality of life among patients experiencing neuropathic pain in the acute inpatient rehabilitation setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have acute or chronic neuropathic pain of any etiology (traumatic, non-traumatic, central, peripheral, and mixed cases).
* Ability to provide informed consent.
* Ability to speak English and complete all aspects of this trial.
* At least 18 years of age.
* Patients will have stable neuropathic pain medication dosing for 3 days prior to enrollment to include gabapentin, pre-gabalin, TCAs, duloxetine, carbamazepine, oxcarbazepine, and venlafaxine).

Exclusion Criteria:

* Patients with platelet count <50,000 or known bleeding disorder.
* Patients in a severe immunocompromised state.
* Pregnant women. All patients who meet the criteria will have their medical records reviewed to ensure they are not pregnant.
* Allergy to gold.
* Use of non-FDA approved herbal supplements. Their effect on enhancing or blunting effect of acupuncture is not known. Patients using medical marijuana with an approved prescription from a state issuing such prescriptions will not be excluded.
* Current infection of the skin or cartilage of the ear.
* Patients already using adjuvant modalities such as chiropractic, massage, yoga, tai chi, massage will not be excluded, but those who add in these modalities during the course of the intervention and observation period will be excluded.
* Patients not anticipated to stay for a minimum of 7 days after enrollment.
* Patient without mental capacity to participate in the consent process and the questionnaire responses.
* Fear of needles or no interest in acupuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported neuropathic pain scores | Daily during inpatient stay, approximately 7-10 days
  Measured on the numeric rating scale for pain (NRS Pain) for pain intensity using a scale of 0=no pain, 10=worst imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Tony Chon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials